CLINICAL TRIAL: NCT04353843
Title: Identification of Clinical, Biometrical and Operatory Factors Related to Pain During Cataract Surgery / RECHMPL20_0210
Brief Title: Identification of Clinical, Biometrical and Operatory Factors Related to Pain During Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other); Beziers Champeau Clinic (Unknown); Montpellier Beau Soleil Clinic (Unknown); Montpellier Ophtalmology Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0210
Record Dates: First submitted 2020-04-17; First posted 2020-04-20 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Cataract
Keywords: Cataract surgery; Phakoemulsification; Pain; Biometry; Anesthesia
MeSH Terms: conditions — Cataract; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adults who undergo cataract surgery will be questioned after surgery about the eventual pain they experienced, about their health history, personal treatment. If they accept to be included in the study we'll record different parameters related to the surgery: type of anesthesia, duration of surgery, machines used, unexpected events, particularities noticed by the surgeon, etc.

There will be no unusual intervention, everything will be run exactly as if there was no study. No additional consultation needed.

DETAILED DESCRIPTION:
Adults who undergo cataract surgery, excepting under general anesthesia, will be asked to rate a Visual Analog Scale grading the pain they experienced, about their health history, personal treatment. If they accept to be included in the study we'll record different parameters related to the surgery: Visual analog scale of pain according to the surgeon (before recording the patient), type of anesthesia, duration of surgery, machines used, time of ultrasound used for phakoemulsification, preoperoative visual acuity and intraocular pressure, biometry, iris color, preoperative donesis, preoperative capsular pseudoexfolliation, unexpected events, particularities noticed by the surgeon as Floppy iris syndrome, Lens-iris diaphragm retropulsion syndrome There will be no unusual intervention, everything will be run exactly as if there was no study. No additional consultation needed.

ELIGIBILITY:
Inclusion criteria:

* Undergoing a cataract surgery during the period of inclusion, and by one of the surgeons of the study
* Majority 18 years and more

Exclusion criteria:

- General anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care population from two clinics and two university hospitals from 3 cities in total, who undergo cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain during cataract surgery | 1 day
  Visual Analog Scale of pain

SECONDARY OUTCOMES:
assess the rate of intraoperative complications over the series | 1 day
  assess the rate of intraoperative complications over the series

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Daien, MD, PhD, HDR, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC